CLINICAL TRIAL: NCT03383705
Title: VBeam Prima for Treatment of Photoaged Facial Skin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DHF24491
Record Dates: First submitted 2017-12-07; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Photoaged Facial Skin
Keywords: Photoaged Skin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment arm (Experimental)
  Interventions: Device: VBeam Prima

INTERVENTIONS:
Device: VBeam Prima — Up to four treatments will be performed every 4-6 (±1) weeks.

SUMMARY:
This is an open-label, single-center study. Subjects in this study will receive up to four (4) facial treatments at 4-6 (±1) weeks interval, with the VBeam Prima device according to the study protocol. Subjects will return for follow-up (FU) visits at the clinic at 1 and 3 months following the last treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Male or Female at least 18 years of age
2. Photoaged facial skin with clinically visible background erythema, telangiectasia, or pigmented lesions
3. Fitzpatrick Elastosis Score 2-9
4. Fitzpatrick Skin Type I - VI
5. Able to read, understand and sign the Informed Consent Form
6. Willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions
7. Willing to have limited sun exposure for the duration of the study, including the follow-up period
8. Willing to have photographs taken of the treated area which will be used, de-identified, in evaluations and may be used, de-identified, in presentations and/or publications
9. For female candidates - subject must be post-menopausal, or surgically sterilized, or using a medically acceptable form of birth control during the entire course of the study.

Exclusion Criteria:

1. Pregnant or planning to become pregnant during the study duration.
2. Implant in the treated area (such as metal plates or screws) or an injected chemical substance.
3. Known collagen (connective tissue) disorder, vascular disease (i.e. saphenous reflux), scleroderma or other autoimmune disease (i.e. rheumatoid arthritis, lupus).
4. History of diseases stimulated by heat or sun exposure, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
5. History of immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
6. Undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including actinic keratosis, presence of malignant or pre-malignant pigmented lesions.
7. Significant concurrent illness, such as such as cardiac disorders, diabetes (type I or II), or pertinent neurological disorders.
8. Infection or are suffering from a current or a history of significant skin conditions in the treated area and/or inflammatory skin conditions, including, but not limited to: photodermatoses, psoriasis, eczema, rash, severe open wound stage rosacea, open cuts or scrapes and active cold sores or herpes sores prior to study treatment or during the study treatment course.
9. Anticoagulative or thromboembolic condition or taking anticoagulation medications one week prior to and during the treatment course (to allow inclusion, temporary cessation of use might be requested as per the subject's physician discretion).
10. Use of aspirin or pain relievers from the ibuprofen family (e.g., Motrin®, Advil®, or Naprosyn®) on a regular basis or would be taking any of these pain relievers one week before and after each study treatment session.
11. History of keloid scarring or of abnormal wound healing.
12. Photosensitivity to the device's laser wavelengths, history of ingesting medications known to induce photosensitivity, or history of seizure disorders due to light.
13. Surgical, light-based therapy or RF procedures in the treatment area within 3 months of treatment or during the study.
14. Any other surgery in the treated area within 3 months of treatment (or more if skin has not healed completely) or during the study.
15. Tattoo or permanent make-up in the treated area.
16. Systemica use of retinoids (i.e. Retin-A®, Accutane®) or antioxidants (i.e. Restylane®, Strivectin®) within 2 months of study treatment or during the study.
17. Excessive tan in areas to be treated or unable/unlikely to refrain from tanning during the study.
18. Participation in a study of another device or drug within three months prior to enrollment or during the study.
19. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-11-15 (Actual); Primary Completion 2018-11-15 (Estimated); Study Completion 2018-11-15 (Estimated)

PRIMARY OUTCOMES:
Global Improvement Scale | 1 or 3 months post last treatment
  Overall improvement using Global Improvement Scale (0=no response; 4=excellent response).

SECONDARY OUTCOMES:
Wrinkle and Elastosis Score | Pre Tx.4, 1 month and 3 months post final treatment
  Improvement using Fitzpatrick Wrinkle Class and Elastosis Score
Treatment discomfort based on NRS Scale | Immediately post treatment
  Evaluate treatment discomfort based on NRS Scale as reported by study subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No